CLINICAL TRIAL: NCT06297525
Title: An Open-Label, Phase 1 Study to Evaluate Safety, Tolerability and Pharmacokinetics of the CTPS1 Inhibitor STP938 in Adult Subjects With Advanced Solid Tumors, With a Safety Expansion in Advanced CTPS2 Null Ovarian Cancer
Brief Title: Study of STP938 in Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Step Pharma, SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STP938-201
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to a dose level of STP938 (Phase 1a) or an expansion cohort (Phase 1b) at the time of their enrollment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a (Part 1, Dose Escalation) (Experimental): Up to 5 dose levels with STP938 administered as oral monotherapy
  Interventions: Drug: STP938
- Phase 1b (Part 2, Safety Expansion) (Experimental): Further evaluation of STP938 administered as oral monotherapy at the RP2D
  Interventions: Drug: STP938

INTERVENTIONS:
Drug: STP938 — Small molecule

SUMMARY:
The Phase 1a part of the study is a dose escalation of STP938 as a monotherapy.

The Phase 1b part of the study is a safety expansion cohort of STP938 as a monotherapy.

ELIGIBILITY:
Main Inclusion Criteria:

* Signed and dated informed consent, and able to comply with the study procedures and any locally required authorization.
* Male or female aged ≥ 18 years.
* Advanced disease not curable by available therapies and requires systemic therapy.
* Histologically confirmed diagnosis of eligible cancer type.
* Must have tumor tissue available for biomarker testing.
* Measurable disease (Part 1) and measurable disease per RECIST (Part2)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Life expectancy > 3 months as assessed by the Investigator.
* Adequate organ function (bone marrow, hepatic, renal function and coagulation).
* All toxicities (except alopecia) from prior cancer treatments or procedures must have resolved to ≤Grade 1 or returned to baseline levels prior to enrollment.

Main Exclusion Criteria:

* Pregnant or breastfeeding females and women of childbearing potential or males unwilling to comply with contraception requirements.
* Known active or symptomatic CNS metastases, carcinomatous meningitis, leptomeningeal disease or a history of spinal cord compression
* Active malignancy within 2 years of study enrollment
* Prior radiation within 2 weeks of start of therapy.
* Systemic cancer treatments, monoclonal antibody-directed therapies, other investigational agents within 4 weeks before enrollment, or <5 half-lives since completion of previous investigational therapy, whichever is shorter.
* Uncontrolled intercurrent illness.
* Immunocompromised subjects with increased risk of opportunistic infections or history of opportunistic infection in the last 12 months.
* Known active or chronic hepatitis B or active hepatitis C virus (HCV) infection.
* Subjects with corrected QT interval >470 msec based on averaged triplicate electrocardiogram (ECG) readings at the Screening Visit using the QT interval corrected for heart rate using Fridericia's method (QTcF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Through study completion, an average of 6 months
  Incidence of dose limiting toxicities (DLTs), serious adverse events (SAEs), treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Area under the curve (AUC) of STP938 | 9 days
  Pharmacokinetic parameter from plasma STP938 levels
Maximum plasma concentration (Cmax) | 9 Days
  Pharmacokinetic parameter from plasma STP938 levels
Time to reach maximum concentration (TMax) | 9 Days
  Pharmacokinetic parameter from plasma STP938 levels
Evaluation of preliminary clinical activity of STP938 | Through study completion, an average of 6 months
  Evaluation of ORR using standard response criteria
Evaluation of best overall response of STP938 | Through study completion, an average of 6 months
  Evaluation of best overall response (Complete response [CR], Partial response [PR], Stable disease [SD], Progression of disease [PD], Not evaluable, Not applicable) using standard response criteria
Evaluation of Duration of Response | Through study completion, an average of 6 months
  Duration of response (DoR) is defined as the time, in days, from the date measurement criteria that are first met for CR or PR (whichever is first recorded) to the first date that relapse, progressive disease or death, whichever occurs first
Evaluation of Progression Free Survival | Through study completion, an average of 6 months
  Progression-free survival (PFS) is defined as the time from first STP938 dose to the date of disease progression or death, whichever occurs first
Change in serum CA125 (ovarian cancer only) | Through study completion, an average of 6 months
  Evaluation of CA125 using standard response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Higgins, Study Director — Step Pharma
Locations (7):
- United States (3):
  - Comprehensive Hematology Oncology, LLC, St. Petersburg, Florida
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Next Oncology, San Antonio, Texas
- Institut Gustave Roussy, Villejuif, Paris, France
- United Kingdom (3):
  - The Beatson Institute for Cancer Research, Glasgow
  - University College London, London
  - The Christie, Manchester